CLINICAL TRIAL: NCT07223359
Title: The Impact of Photographic Evidence on Postoperative Range of Motion Following Total Knee Arthroplasty: A Randomized Control Trial
Brief Title: Photographic Evidence on Total Knee Arthroplasty Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Nicholas Brown, Principal Investigator, Loyola University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LU213164
Record Dates: First submitted 2025-10-27; First posted 2025-10-31 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Osteoarthritis (OA) of the Knee
Keywords: total knee arthroplasty; range of motion; photographic outcomes
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Photographic Evidence Group (Experimental): Participants in this group will receive printed photographs of their operated knee in full flexion and full extension immediately following total knee arthroplasty (TKA). The photographs will be taken in the operating room after dressings are applied. Patients will be instructed to keep one copy for personal use and to provide another copy to their physical therapist. The goal of this intervention is to determine whether visual feedback of postoperative range of motion enhances motivation, engagement in rehabilitation, and early recovery.
  Interventions: Behavioral: Photographic Evidence of Postoperative Knee Range of Motion
- Control Group (Active Comparator): Participants in this group will undergo total knee arthroplasty (TKA) and receive standard postoperative management and rehabilitation without photographs of their knee range of motion. They will participate in the same physical therapy and follow-up schedule as the intervention group.
  Interventions: Behavioral: Standard Postoperative Care

INTERVENTIONS:
Behavioral: Photographic Evidence of Postoperative Knee Range of Motion — The intervention consists of providing patients with photographic evidence of their knee range of motion (ROM) immediately following total knee arthroplasty (TKA). After the procedure, while still in the operating room and after sterile dressings are applied, two photographs are taken of the operated knee, one in maximum flexion and one in full extension.
  Arms: Photographic Evidence Group
Behavioral: Standard Postoperative Care — Participants will receive routine postoperative management and physical therapy following TKA. No photographic evidence of knee range of motion will be provided.
  Arms: Control Group

SUMMARY:
Historically, total knee arthroplasty (TKA) has been performed to restore knee range of motion and relieve pain, with postoperative rehabilitation focused on helping patients regain mobility and function. This study evaluates whether providing patients with photographic evidence of their knee range of motion immediately after surgery can enhance short-term recovery.

Patients will be randomly assigned to one of two groups: one group will receive printed photographs showing their knee in full flexion immediately after surgery, while the other group will not receive photographs. Outcomes assessed at six weeks postoperatively will include knee range of motion, physical therapy progress metrics, length of hospital stay, and patient-reported outcomes.

DETAILED DESCRIPTION:
Participants include patients 18 years or older presenting to the investigators' institutions who are scheduled to undergo a primary total knee arthroplasty (TKA). Exclusion criteria include revision TKA, prior surgery or fracture involving the operative knee, preoperative knee flexion contracture greater than 10 degrees, patients with comorbidities, and those unable or unwilling to provide informed consent.

If, after evaluation, the patient remains eligible, the surgeon will introduce the study. If the patient expresses interest, a member of the study team will approach the patient to explain the study in detail. The voluntary nature of participation will be emphasized, and the prospective participant will be encouraged to ask questions and discuss participation with others. Once all questions have been addressed, the participant will be presented with the informed consent document (ICD). The study team member will step out of the room to allow time for review. If desired, the participant may take a paper copy of the ICD to discuss with family or others before signing. Once all questions have been answered to the participant's satisfaction, the ICD will be signed, preferably in the clinic. If the participant elects to take the ICD home, a follow-up time will be arranged, typically during preoperative clearance or on the day of surgery to review and sign the document.

After informed consent is obtained, preoperative baseline data including range of motion and patient-reported outcome measures will be collected. Participants will then be randomized in a 1:1 fashion to either receive or not receive photographic evidence of their postoperative knee range of motion. Randomization will be performed using stratified randomization lists generated and maintained by the Biostatistics Core at Loyola University Clinical Research Office to ensure equal allocation across sites.

During surgery, photographs of the operated knee in full flexion and full extension will be taken. Participants randomized to the intervention group will receive printed copies of the photographs and instructions to share them with their physical therapist. The control group will not receive any photographs. All participants will receive standard perioperative management, surgical technique, and rehabilitation protocols.

The primary outcome is knee flexion at six weeks postoperatively, measured using a goniometer by a blinded assessor. Secondary outcomes include knee extension, physical therapy progress metrics (total duration of therapy, time to achieve 110 degrees of flexion, and number of therapy sessions), distance walked on postoperative day one, length of hospital stay, and patient-reported outcomes via the Knee Injury and Osteoarthritis Outcome Score (KOOS) survey.

A sample size of 52 patients (26 per group) was calculated to provide 80% power to detect a 10-degree difference in knee flexion at six weeks, assuming a standard deviation of 12 degrees and a two-sided alpha level of 0.05.

Both groups will undergo standard postoperative follow-up at two weeks, six weeks, and as per routine care thereafter. Data collection at each time point will include range of motion assessments, physical therapy metrics, and KOOS surveys.

The investigators hypothesize that providing photographic evidence of postoperative knee range of motion will enhance patient motivation and engagement in rehabilitation, resulting in improved early range of motion and functional recovery compared to standard rehabilitation alone.

Participation in this study carries minimal risk. All procedures, surgical techniques, and follow-up care are consistent with the standard of care for patients undergoing TKA. The primary risk to participants is potential loss of confidentiality, which is rare. There are no additional surgical risks associated with participation. Subject safety will be monitored during routine postoperative visits, and participants will have access to the study team for any questions or concerns.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Scheduled to undergo primary unilateral total knee arthroplasty (TKA) at one of the investigators' participating institutions
* Able to understand study procedures and comply with follow-up requirements
* Able to read and complete questionnaires in English
* Willing and able to provide informed consent prior to participation

Exclusion Criteria:

* Undergoing revision TKA
* History of prior surgery or fracture involving the operative knee
* Preoperative knee flexion contracture >10 degrees
* Patients with non-elective or trauma-related indications for knee replacement
* Inability or unwillingness to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Knee Flexion at Six Weeks Postoperatively | 6 weeks after total knee arthroplasty
  Knee flexion will be measured in degrees using a goniometer by a blinded assessor at the 6-week postoperative visit. The outcome compares the degree of maximum flexion between participants who received photographic evidence of their postoperative range of motion and those who did not.

SECONDARY OUTCOMES:
Knee Extension at Six Weeks Postoperatively | 6 weeks after total knee arthroplasty
  Knee extension will be measured in degrees using a goniometer by a blinded assessor at the 6-week postoperative visit.
Total Duration of Physical Therapy | Up to 6 weeks after surgery
  Total duration of physical therapy from initiation to completion, measured in weeks, as documented in the medical record.
Length of Hospital Stay | From the date of surgery until the date of hospital discharge, assessed for up to 6 weeks postoperatively.
  Length of stay (LOS) will be measured as the number of days from the date of surgery to the date of hospital discharge.
Total Number of Physical Therapy Sessions | Up to 6 weeks after surgery
  Total number of in-person physical therapy sessions completed during the postoperative period, as documented in the medical record.
Time to Achieve 110° of Knee Flexion (Weeks) | Up to 6 weeks after surgery
  Number of weeks from surgery until the patient achieves 110° of knee flexion during physical therapy, as documented in the medical record.
Time to Achieve 110° of Knee Flexion (Sessions) | Up to 6 weeks after surgery
  Number of physical therapy sessions required for the patient to achieve 110° of knee flexion, as recorded in the physical therapy documentation.
Distance Walked on Postoperative Day One | Postoperative day 1
  Distance walked during the first postoperative physical therapy session, measured in feet, as documented in the physical therapy record.
Patient-Reported Outcome Measures (KOOS Survey) | 6 weeks after surgery
  Patient-reported outcomes will be measured using the Knee Injury and Osteoarthritis Outcome Score (KOOS) survey, a validated instrument assessing five subscales: Pain, Symptoms, Activities of Daily Living (ADL), Sports and Recreation Function, and Knee-Related Quality of Life (QOL).
  Each subscale is scored from 0 to 100, where 0 represents extreme knee problems and 100 represents no knee problems.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Loyola University Medical Center, Maywood, Illinois
  - Gottlieb Memorial Hospital, Melrose Park, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roos EM, Lohmander LS. The Knee injury and Osteoarthritis Outcome Score (KOOS): from joint injury to osteoarthritis. Health Qual Life Outcomes. 2003 Nov 3;1:64. doi: 10.1186/1477-7525-1-64. PMID 14613558
- [Background] Abson S, Kenny B, Rahim R, Benz D, Hellman J. Can visual aides influence rehabilitation and length of stay following knee replacement? A randomized controlled study. Orthop Rev (Pavia). 2015 Mar 31;7(1):5758. doi: 10.4081/or.2015.5758. eCollection 2015 Mar 3. PMID 25874065
- [Background] Pinsornsak P, Kanitnate S, Boontanapibul K. The effect of immediate post-operative knee range of motion photographs on post-operative range of motion after total knee arthroplasty : An assessor-blinded randomized controlled clinical trial in sixty patients. Int Orthop. 2021 Jan;45(1):101-107. doi: 10.1007/s00264-020-04877-3. Epub 2020 Nov 24. PMID 33230607
- [Background] Farahini H, Moghtadaei M, Bagheri A, Akbarian E. Factors influencing range of motion after total knee arthroplasty. Iran Red Crescent Med J. 2012 Jul;14(7):417-21. Epub 2012 Jul 30. PMID 22997557
- [Background] Hyodo K, Masuda T, Aizawa J, Jinno T, Morita S. Hip, knee, and ankle kinematics during activities of daily living: a cross-sectional study. Braz J Phys Ther. 2017 May-Jun;21(3):159-166. doi: 10.1016/j.bjpt.2017.03.012. Epub 2017 Apr 9. PMID 28473283
- [Background] Laubenthal KN, Smidt GL, Kettelkamp DB. A quantitative analysis of knee motion during activities of daily living. Phys Ther. 1972 Jan;52(1):34-43. doi: 10.1093/ptj/52.1.34. No abstract available. PMID 5061683